CLINICAL TRIAL: NCT01377155
Title: A Comparison of Two Initial Dosing Formulas for Basal Insulin in Type 2 Diabetes Mellitus
Brief Title: A Comparison of Two Initial Dosing Formulas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diabetes Care Center (Industry)
Responsible Party: Principal Investigator, Allen B. King, MD, Principal Investigator, Diabetes Care Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DCC 03-11
Record Dates: First submitted 2011-06-17; First posted 2011-06-21 (Estimated); Last update posted 2013-08-27 (Estimated); Status verified 2013-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: basal insulin; hypoglycemia; diabetes mellitus type two
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypoglycemia | interventions — Insulin Detemir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Insulin determir (Other)
  Interventions: Drug: Insulin detemir

INTERVENTIONS:
Drug: Insulin detemir — Subjects will be randomized to weight based method of 0.1 U/kg for basal insulin or a starting dose based upon an insulin challenge. Subject will record morning fasting blood sugar daily. Using a three day average, the subject will titrate the dose of basal insulin either increasing or lowering by three units based upon target blood glucose of 110 mg/dl.

SUMMARY:
This study will evaluate two methods of starting basal insulin to see which method may achieve a faster-to-goal titration.

DETAILED DESCRIPTION:
The current recommended starting dose of basal insulin in type 2 diabetes is either a fixed dose, e.g. 10 U, or a weight-based formulas, 0.1-0.2 U/kg. The estimate of eventual titration dose to attempt to reach a fasting glucose goal is 0.49 U/kg. Those many weeks of dosage upward titration are required. The investigators propose to compare the current recommended weight based, 0.1 U/kg to a correction factor derived formula. Starting with an insulin tolerance test estimation of basal dose, one would arrive at the eventual titrated basal insulin dose in significantly less days than starting at a starting dose estimate of 0.1 U/kg. Further, there would be no significant increase in overall reported hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes
2. Age 18 years and above
3. Concurrently on ± sulfonylureas ± thiazolidinedione ± DDP IV inhibitors ± metformin ± glinides
4. A1c ≥ 7.0% but ≤ 10%
5. Capable of self monitoring glucose ≥4/day
6. Previously compliant with clinical recommendations
7. Fasting blood glucose ≥ 150 mg/dl
8. BMI ≤ 45 kg/m2

Exclusion Criteria:

1. Urinary ketosis
2. Currently or expected alteration in insulin sensitivity such as major surgery, infection, renal failure (creatinine >1.5 mg/dl), glucocorticoid treatment, recent (within 2 weeks) serious hypoglycaemic episode (requires assistant of another)
3. Currently participating in another clinical trial
4. Known or suspected allergy to insulin determir
5. Using insulin
6. Pregnancy or nursing or the intention of becoming pregnant or not using adequate
7. Significant liver or heart failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Days to reach the titration target | 12 weeks
  The number of days for the subject to reach the titration target blood sugar of 110 ml/dl

SECONDARY OUTCOMES:
The frequency of reported and documented (<70 mg/dl) hypoglycemic events per 24 hour period | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Allen B King, MD, Principal Investigator — Diabetes Care Center
Locations (1):
- Diabetes Care Center, Salinas, California, United States